CLINICAL TRIAL: NCT05870033
Title: Gender Difference of Muscle Activation Amongst Patients With Knee Osteoarthritis
Brief Title: Muscle Activation in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: Muscle activation
Record Dates: First submitted 2023-05-02; First posted 2023-05-23 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electromyography; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men group: Muscle activity amongst men with KOA
  Interventions: Device: Electromyography (EMG) measurement
- Women group: Muscle activity amongst women with KOA
  Interventions: Device: Electromyography (EMG) measurement

INTERVENTIONS:
Device: Electromyography (EMG) measurement — Electromyography (EMG) measurement of m. quadriceps femoris and semitendinosus muscle during static functional tasks

SUMMARY:
Muscle activity, as a possible fundamental cause of functional limitation, has been extensively investigated in knee osteoarthritis (KOA). Many trials investigated muscle activity during dynamic movements and functional tasks in KOA. In addition, gender-related differences has been also investigated during functional movements in KOA. However, no trial investigated gender-related differences in muscle activation during static movement in KOA.

DETAILED DESCRIPTION:
Muscle activity, as a possible fundamental cause of functional limitation, has been extensively investigated in knee osteoarthritis (KOA). Interestingly, studies concentrated mainly on investigation of muscle activity during dynamic movements and different functional tests. Moznuzzaman et al displayed greater muscle activation during sitting to standing test (STS) and standing to sitting test in KOA patients compared to healthy participants. Interestingly, some studies investigated muscle activation standing up from a knee-height seat during STS and illustrated a greater muscle activation amongst KOA patients compared to healthy controls. Moreover, Amer et al found greater muscle activation while performing STS from a lower height seat compared to a knee-height seat amongst women and men patients with uni/bilateral KOA. These findings might be of interest due to compensatory mechanisms observed by female patients during STS transition increases loading on the joint surfaces and consequently leading to progression of KOA. Furthermore, different studies also presented gender-differences of muscle activation during different weight-bearing tasks (gait, STS, stair ascend/descend, and squat) amongst patients with KOA and healthy control. Interestingly, both studies showed women with KOA representing higher muscle activation compared to men. Therefore, an analytical comparative study might be useful for identification of gender-differences in muscle activation amongst patients with KOA.

Investigation of static muscle activity during functional movements is very rare in KOA. Zhang et al investigated muscle activation after single whole body vibration trial in standing position at 0°, 30° and 60° static knee flexion angles amongst women with KOA. Authors found that muscle activation in 60° was greater compared to 30°, and it was also greater in 30° compared to 0°. Based on our literature search, no further study examined muscle activity in static knee flexion in KOA. However, investigating static knee flexion might be useful as it could be related to different knee moments in KOA.

ELIGIBILITY:
Inclusion Criteria:

* radiologically diagnosed KOA based on the Kellgren-Lawrence grading system 1-3,
* age above 60 years
* at least 60° active knee flexion
* sufficient mental status

Exclusion Criteria:

* acute inflammation of the knee
* intraarticular injections within the last 3 months
* total knee replacement in the opposite side
* class II obesity (body mass index, BMI>35kg/m2)
* severe degenerative lumbar spine disease (e.g., spondylolisthesis)
* systemic inflammatory arthritic or neurological condition
* conservative intervention attendance within 6 months
* contraindication to conservative therapy and manual therapy
* unstable heart condition
* complex regional pain syndrome

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiologically diagnosed KOA
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Patients' baseline state | within 1 day
  Measurement of patients' pain, stiffness and functional state based on WOMAC
Patients' baseline pain | within 1 day
  Measurement of patients' pain based on Numeric Pain Rating Scale
Patients' baseline knee flexion | within 1 day
  Measurement of patients' active knee flexion in supine
Patients' baseline knee flexion in standing position | within 1 day
  Measurement of patients' active knee flexion during weight-bearing
Muscle strength of m. quadriceps femoris | within 1 day
  Measurement of muscle strength of m. quadriceps femoris in 0, 35 and 60 degree
Muscle strength of hamstring muscles | within 1 day
  Measurement of muscle strength of m. semitendinosus, semimembranosus and biceps femoris in 0, 35 and 60 degree
Muscle activation in 30 degree static knee flexion | within 1 day
  EMG measurement of muscle activation during 2-leg 30 degree static knee flexion
Muscle activation in 60 degree static knee flexion | within 1 day
  EMG measurement of muscle activation during 2-leg 60 degree static knee flexion
Muscle activation during stepping up a stair | within 1 day
  EMG measurement of muscle activation during stepping up on a stair
Muscle activation during stepping down a stair | within 1 day
  EMG measurement of muscle activation during stepping down from a stair
Muscle activation during stepping down side-ways a stair with affected leg | within 1 day
  EMG measurement of muscle activation during stepping down side-ways a stair with affected leg
Muscle activation during stepping down side-ways a stair with opposite leg | within 1 day
  EMG measurement of muscle activation during stepping down side-ways a stair with opposite leg
Muscle activation in one-leg standing position | within 1 day
  EMG measurement of muscle activation in one-leg standing position

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Melczer, Physiother., Study Director — University of Pecs
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Amer HS, Sabbahi MA, Alrowayeh HN, Bryan WJ, Olson SL. Electromyographic activity of quadriceps muscle during sit-to-stand in patients with unilateral knee osteoarthritis. BMC Res Notes. 2018 Jun 5;11(1):356. doi: 10.1186/s13104-018-3464-9. PMID 29871669
- [Background] Bouchouras G, Sofianidis G, Patsika G, Kellis E, Hatzitaki V. Women with knee osteoarthritis increase knee muscle co-contraction to perform stand to sit. Aging Clin Exp Res. 2020 Apr;32(4):655-662. doi: 10.1007/s40520-019-01245-z. Epub 2019 Jun 15. PMID 31203528
- [Background] Smith SL, Woodburn J, Steultjens MPM. Sex- and osteoarthritis-related differences in muscle co-activation during weight-bearing tasks. Gait Posture. 2020 Jun;79:117-125. doi: 10.1016/j.gaitpost.2020.04.019. Epub 2020 Apr 27. PMID 32402893